CLINICAL TRIAL: NCT00271128
Title: NT-proBNP for Evaluation of the Dyspneic Patient in the Emergency Room and the Medical Ward (BNP4EVER)
Brief Title: NT-proBNP for Evaluation of the Dyspneic Patient in the Emergency Room and the Medical Ward
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: hymc34/2005
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2005-12

CONDITIONS: Shortness of Breath; Acute Exacerbation
Keywords: NT-proBNP; Heart failure; Dyspnea
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The proposed study intends to evaluate the impact of the NT-proBNP assay on the diagnosis of heart failure in patients with dyspnea of unknown etiology presenting to the emergency room and admitted to the medical wards.

DETAILED DESCRIPTION:
The proposed study intends to evaluate the impact of the NT-proBNP assay on the diagnosis of heart failure in patients with dyspnea of unknown etiology presenting to the emergency room and admitted to the medical wards.

Patients will be consented and randomized to open or blinded NT-proBNP test performed within 90 minutes in a venous blood sample.

Evaluation of the ER diagnosis and final discharge diagnosis in admitted patients will be carried out in light of the NT-proBNP results.

ELIGIBILITY:
Inclusion Criteria:

1. Acute shortness of breath of unknown etiology as presentation to the emergency room
2. Possible acute exacerbation of known heart failure

Exclusion Criteria:

None -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-10; Study Completion 2007-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Simcha R Meisel, MD MSc, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Meisel SR, Januzzi JL, Medvedovski M, Sharist M, Shochat M, Ashkar J, Peschansky P, Haim SB, Blondheim DS, Glikson M, Shotan A. Pre-admission NT-proBNP improves diagnostic yield and risk stratification - the NT-proBNP for EValuation of dyspnoeic patients in the Emergency Room and hospital (BNP4EVER) study. Eur Heart J Acute Cardiovasc Care. 2012 Jun;1(2):99-108. doi: 10.1177/2048872612447049. PMID 24062895